CLINICAL TRIAL: NCT05205850
Title: An Open, Multi-center Phase I/IIa Clinical Study of RC118 for Injection in Patients with Locally Advanced Unresectable or Metastatic Malignant Solid Tumors with Positive Expression of Claudin 18.2
Brief Title: A Study of RC118 in Patients with Locally Advanced Unresectable or Metastatic Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC118-C001
Record Dates: First submitted 2021-11-17; First posted 2022-01-25 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC118-ADC (Experimental): Participants will be allocated to one of the following dose groups: 0.25, 0.5, 1.0, 1.5, 2.0, 2.5, and 3.0mg/kg, and receive a treatment of RC118-ADC followed by 14 days of dose limited toxicity (DLT) observation period.
  Interventions: Drug: RC118-ADC

INTERVENTIONS:
Drug: RC118-ADC — RC118 for injection is a novel antibody-drug conjugate, with a Claudin 18.2-targeting antibody and a microtube inhibitor
  Other Names: RC118 for injection

SUMMARY:
In Phase I, This study will explore the tolerability and safety of RC118 in patients with locally advanced unresectable or metastatic malignant solid tumors with positive Claudin 18.2 expression, and determine the maximum tolerated dose (MTD) and the recommended dose in phase II clinical trials (RP2D); In Phase IIa, to explore the clinical effectiveness and safety of long-term use of RC118 at RP2D doses for patients with different tumor types。

DETAILED DESCRIPTION:
this study is an open, single arm, multi-center Phase I /IIa clinical study. In the phase I, patients with locally advanced unresectable or metastatic malignant solid tumors (gastric cancer, esophageal cancer, gastroesophageal junction cancer, pancreatic cancer, ovarian cancer, cholangiocarcinoma, etc.) that are positive for Claudin 18.2(positive membrane staining observed in any tumor cells) will be included. in Phase I dose escalation phase, 7 dose groups will be preset：0.25 mg/kg、0.5 mg/kg、1.0 mg/kg、1.5 mg/kg、2.0 mg/kg、2.5 mg/kg、3.0mg/kg; In phase I dose confirmation phase, it is initially considered to set up 1~2 dose groups according to the dose-escalation phase MTD/MAD, with 3~6 subjects in each group. In the phase IIa cohort expansion phase, with reference to the results of the phase I study, subjects were grouped according to different tumor types, there are 30 subjects in each group, initially considering the inclusion of Claudin 18.2 positive(a clear cut-off value will be defined based on the results of Phase I) locally advanced unresectable or metastatic gastric cancer, esophageal cancer, gastroesophageal junction cancer, and pancreatic cancer patients.(The specific tumor types and groups will be further adjusted based on the results of the phase I study).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study and sign written informed consent
2. 18 years old ≤ age ≤ 75 years old, no gender limit
3. ECOG physical status score is 0 or 1 point
4. The expected survival time exceeds 12 weeks
5. Standard treatment is ineffective (disease progression or no remission after treatment), patients who cannot tolerate standard treatment, locally advanced unresectable or metastatic malignant solid tumors
6. The subject agrees to provide freshly collected tumor tissue specimens or collected and preserved tumor tissue specimens within 2 years during the screening period for CLDN 18.2 testing, and must meet the following criteria： A.Phase I dose escalation stage/dose confirmation stage: patients with gastric cancer, esophageal cancer, gastroesophageal junction cancer, pancreatic cancer, ovarian cancer, and cholangiocarcinoma with positive Claudin 18.2 expression (membrane staining is observed in any tumor cells); B.Phase IIa Dose Expansion phase: (positive membrane staining observed in any tumour cell) patients with gastric/gastro-oesophageal adenocarcinoma, pancreatic cancer; C. Phase IIa dose-optimisation phase: patients with gastric/gastro-oesophageal adenocarcinoma with Claudin 18.2-positive (positive membrane staining observed in any tumour cell)
7. According to the RECIST v1.1 standard, based on imaging examination (CT/MRI), there is at least one measurable or evaluable target lesion
8. Sufficient bone marrow, liver, and kidney functions (subject to the normal value of the clinical trial center): absolute neutrophil count (ANC) ≥ 1.5×109/L, platelet ≥ 100×109/L, hemoglobin ≥ 90 g/ L, serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN), ALT, AST or ALP ≤ 3 times ULN without liver metastasis; ALT, AST or ALP ≤ 5 times ULN with liver metastasis, serum creatinine ≤ 1.5 Times ULN, International Normalized Ratio (INR) ≤ 1.5 times ULN, APTT ≤ 1.5 times ULN
9. Male or female subjects with fertility must agree to take effective contraceptive measures during the study period and within 6 months after the end of the last medication, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or women whose blood pregnancy test results are positive during the screening period (female subjects who are infertile do not need to undergo a pregnancy test, such as hysterectomy and/or bilateral ovaries in the past Women with resection or amenorrhea ≥12 months)
2. Subjects with positive test results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), and human immunodeficiency virus antibody (HIV-Ab) during the screening period
3. Subjects with a prior history of other acquired, congenital immunodeficiency diseases; subjects who are preparing for or have previously undergone organ or bone marrow transplantation;
4. Those who have previously received targeted therapy drugs for Claudin 18.2; or participated in clinical trials of other drugs within 4 weeks before the first administration and received trial drugs
5. Have vaccinated within 4 weeks before the first dose or plan to vaccinate any vaccine during the study period
6. Allergic to known research drug ingredients or excipients
7. Combined use of vitamin K antagonist anticoagulant drugs; combined use of therapeutic doses of heparin (subjects using preventive doses of heparin can be included in the study)
8. Received anti-tumor therapy (surgery, chemotherapy, radiotherapy, biological therapy) within 4 weeks before the first administration, and received palliative radiotherapy for bone metastases within 2 weeks
9. The toxicity of previous anti-tumor treatments has not returned to the level 0 or 1 of NCI-CTCAE v5.0 (except for hair loss)
10. There are clinical symptoms of pleural fluid, ascites, and pericardial effusions require drainage (patients who do not require drainage or whose drainage is discontinued and who do not have a significant increase in effusion within 5 days may be included in the study)
11. According to the judgment of the investigator, an active infection with clinical significance
12. Combined with other diseases that seriously endanger the safety of the subject or affect the completion of the test, such as gastrointestinal bleeding (within 4 weeks before the first dose), peptic ulcer, intestinal obstruction, intestinal paralysis, interstitial pneumonia, lung Fibrosis, kidney failure, and uncontrolled diabetes
13. QTc interval during the screening period>480 ms (based on the average of 3 screening electrocardiograms); previous family or personal history of long/short QT interval syndrome; ventricular arrhythmia deemed clinically significant by the investigator Medical history, or currently receiving antiarrhythmic drug treatment, or implantation of arrhythmia defibrillation device
14. Past myocardial infarction (within 6 months before the first administration), severe or unstable angina, coronary or peripheral artery bypass grafting, New York Heart Association (NYHA) grade 3~4 heart failure, no Controlled hypertension
15. People who have had alcohol dependence or drug abuse in the past
16. Those who have received systemic steroid therapy for a long period of time (Note: Short-term use (≤ 7 days) and withdrawal> 2 weeks can be selected)
17. Patients who have previously or currently suffered from uncontrolled primary or metastatic brain tumors, and the investigator believes that patients who have been stabilized or whose local treatment has ended may be considered for inclusion in the group
18. Past or current peripheral neuropathy ≥ Grade 2
19. Past or current mental illness that is difficult to control
20. Subjects who have poor compliance and are not expected to cooperate to complete the test procedure
21. Other subjects deemed unsuitable to participate in clinical research by the investigator
22. Serious arterial/venous thrombosis or cardiovascular accident within 6 months prior to dose administration, such pulmonary embolism, cerebral infarction, cerebral hemorrhage, except for asymptomatic lacunar infarction that does not require clinical intervention;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days after first treatment.
  In the DLT evaluation window (observation period 1-28 days after the first administration), according to the NCI-CTCAE v5.0 grading standard, the investigator or the sponsor believes that toxic reaction which are reasonably related to RC118 treatment
The incidence and severity of adverse events (AE) | From the day of ICF sign to 28 days after the day of the last treatment
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v5.0
Objective response rate (ORR) | 15 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 15 months
  Disease Control Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR) or stable disease(SD)
Progression-free survival (PFS) | 15 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Duration of Remission (DOR) | 15 months
  Duration of response is the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Pharmacokinetic index | 15 months
  Tmax ，etc.
Immunogenicity | 15 months
  Anti-drug antibody (ADA) positive samples, etc.
Overall survival（OS） | Up to approximately 2 years
  OS was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tianshu Liu, ph.D, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The first affiliated hospital, zhejiang universtity school of medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No